CLINICAL TRIAL: NCT03224780
Title: Creatine Kinase Versus 3D Doppler for Antenatal Diagnosis of Morbidly Adherent Placenta
Brief Title: Creatine Kinase Versus 3D Doppler for Antenatal Diagnosis of Abnormal Adherent Placenta.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Nesreen Abdel Fattah Abdullah Shehata, Assistant Professor of Obstetrics and Gynecology, Beni-Suef University
Other Study IDs: Beni-Suef 13
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: maternal serum creatine kinase — Biochemical marker
Diagnostic Test: 3D Doppler ultrasound — Doppler for placental vessels

SUMMARY:
Placenta accreta is a potentially life-threatening obstetric condition that requires a multidisciplinary approach to management.Diagnosis of placenta accreta before delivery minimizes potential maternal or neonatal morbidity and mortality. In this study the researchers will evaluate the role and cost effectiveness of biochemical marker as creatine kinase in comparison with 3D Doppler ultrasound in antenatal diagnosis of placenta accreta and its variants in patients with placenta previa totalis.

DETAILED DESCRIPTION:
Abnormal placentation poses a diagnostic and treatment challenge for all providers caring for pregnant women. As one of the leading causes of postpartum hemorrhage, abnormal placentation involves the attachment of placental villi directly to the myometrium with potentially deeper invasion into the uterine wall or surrounding organs. Surgical procedures that disrupt the integrity of uterus, including cesarean section, dilatation and curettage, and myomectomy, have been implicated as key risk factors for placenta accreta(Megier et al., 2000).Prenatal diagnoses of placenta accreta through the use of gray-scale ultrasonography, color Doppler imaging, and magnetic resonance imaging have been reported previously (Chou et al., 1997).

Placenta increta and percreta have rarely been diagnosed antepartum, and ultrasonographic findings may provide the only objective evidence of placenta accreta.A biochemical marker for this condition would therefore be useful (Ophir et al., 1999).It is critical to make the diagnosis before delivery because preoperative planning can significantly decrease blood loss and avoid substantial morbidity associated with placenta accreta (Shih et al., 2009).

ELIGIBILITY:
Inclusion Criteria:

- a- Pregnant lady with history of previous cesarean section or hysterotomy. b- Placenta previa with its lower edge covering the scar of previous cesarean section as diagnosed by 2DU/S.

c- Gestational age ranging from 28 wks - Full term.

Exclusion Criteria:

* Women with one or more of the following conditions contributing to rhabdomyolysis:

  1. Crush injury and prolonged surgery.
  2. Embolism, thrombosis, D.V.T., myocardial or brain infarction.
  3. Drug overdose: Antipsychotics, antidepressants, hypnotics, narcotics, alcohol, halothane,salicylates.
  4. Excessive muscle activity as epileptic fit.
  5. Chronic hypertension & PIH
  6. Endocrine disorders: hyper-/hypothyroidism, and diabetes mellitus,history of liver disease or renal disease.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnant women with persistent placenta previa (after 28 weeks' gestation) were prospectively enrolled into this study.complete imaging using all diagnostic techniques (gray-scale, color Doppler and 3D power Doppler), and full availability of delivery information. Ultrasound examination was performed using a 3D ultrasound system equipped with a 4-8-MHz transabdominal transducer .• Serum Creatine kinase assessement (reference range is 25-160 U/L).(Ophir et al 1999)
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
maternal morbidity | from 28 weeks gestation until 24 hours postpartum.
  Antepartum and Postpartum maternal complications of morbidly adherent placenta.

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-Suef University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chou MM, Ho ES. Prenatal diagnosis of placenta previa accreta with power amplitude ultrasonic angiography. Am J Obstet Gynecol. 1997 Dec;177(6):1523-5. doi: 10.1016/s0002-9378(97)70102-9. PMID 9423762
- [Background] Megier P, Harmas A, Mesnard L, Esperandieu OL, Desroches A. Picture of the month. Antenatal diagnosis of placenta percreta using gray-scale ultrasonography, color and pulsed Doppler imaging. Ultrasound Obstet Gynecol. 2000 Mar;15(3):268. doi: 10.1046/j.1469-0705.2000.00083.x. No abstract available. PMID 10846790
- [Background] Ophir E, Tendler R, Odeh M, Khouri S, Oettinger M. Creatine kinase as a biochemical marker in diagnosis of placenta increta and percreta. Am J Obstet Gynecol. 1999 Apr;180(4):1039-40. doi: 10.1016/s0002-9378(99)70683-6. PMID 10203680